CLINICAL TRIAL: NCT05048576
Title: The Effect of Auditory Cues on Mood and Gait
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clarkson University (Other)
Responsible Party: Principal Investigator, Ali Boolani, Associate Professor, Clarkson University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-20.2
Record Dates: First submitted 2021-08-13; First posted 2021-09-17 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Psychological; Auditory Perception
MeSH Terms: interventions — SIR1 protein, S cerevisiae; Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Positive auditory cues (Experimental): Participants will listen to the following auditory cues ~30 seconds apart Good job, you're doing awesome! Keep up the good work! You've got this! You're almost done, just a few more minutes! That's a great pace! You're going strong! Keep it up! Nice work. Great job! Good stuff. Keep it up. You're doing an amazing job.
  Interventions: Behavioral: Positive Reinforcement
- Negative auditory cues (Experimental): Participants will listen to the following auditory cues ~30 seconds apart You've got to walk faster than that. You're so slow! Why do you walk like that? Did you learn how to walk yesterday? You're doing terrible. Who walks like that? You have potential but you don't use it. You'll never amount to anything. You're not putting very much effort into this. This is the worst pace you've had yet.
  Interventions: Behavioral: Negative Reinforcement
- Music (Experimental): Participants will be allowed to select a streaming music station of their choice.
  Interventions: Behavioral: Music
- Silence (Active Comparator): Participants will walk in silence while wearing noise cancelling headphones.
  Interventions: Behavioral: Silence

INTERVENTIONS:
Behavioral: Negative Reinforcement — Terms to be used in negative reinforcement:
  You've got to walk faster than that. You're so slow! Why do you walk like that? Did you learn how to walk yesterday? You're doing terrible. Who walks like that? You have potential but you don't use it. You'll never amount to anything. You're not putting very much effort into this. This is the worst pace you've had yet.
  Arms: Negative auditory cues
Behavioral: Positive Reinforcement — Terms to be used in positive reinforcement:
  Good job, you're doing awesome! Keep up the good work! You've got this! You're almost done, just a few more minutes! That's a great pace! You're going strong! Keep it up! Nice work. Great job! Good stuff. Keep it up. You're doing an amazing job.
  Arms: Positive auditory cues
Behavioral: Silence — No recordings will be played during this condition.
  Arms: Silence
Behavioral: Music — Participant's can choose their own music to play during this condition.
  Arms: Music

SUMMARY:
The objective of this study is to identify the influence of positive and negative auditory cues, music and a placebo (silence) on mood and gait during 30 minutes of free walking. Participants will be required to walk for a total of 30 minutes with mood being measured every 5 minutes and gait measured throughout the 30 minute protocol.

ELIGIBILITY:
Inclusion criteria:

* Able to stand without an assistive device

  * This study requires subjects to stand and to walk with the Delsys monitors, thus we are unable to use subjects who cannot stand without assistive devices.
  * Delsys monitors are a wearable device that allows for comprehensive analysis of gait and balance. The sensors will be attached to the subject and they will be instructed to perform the gait test by walking for 5 minute intervals over the duration of 63 minutes. The Delsys will generate a report automatically that will then be analyzed.
* Able to walk in 5-minute intervals over the duration of 63 minutes without assistive devices.

  * The objective of this study is to measure gait. Assistive devices change gait and limit our ability to measure gait.

    • Subjects must be within the age of 18-45

Exclusion criteria:

* Impairment or inability to perform physical activity (e.g. walking) independently.
* Inability to walk for 2 minutes without pain or discomfort.
* Neurological conditions (i.e. stroke or Parkinson's disease)

  ○ Many neurological conditions can potentially alter gait. Therefore, we are eliminating individuals in this group.
* Recent (within 6 months) orthopedic surgery that impacts walking ability and balance, e.g. total joint replacement

  ○ The objective of this study is to measure gait and people with lower extremity injuries may have excessive variation in gait. Hence we will be eliminating them from this study.
* Wound or absent sensation on plantar surface (bottom) of the subject's feet.

  ○ Subjects with this issue will have alterations and variations in gait due to sensory deficits and/or pain. They will not eligible for this study.
* Visual Impairment ○ Subjects must be able to read and visually recognize words. Therefore, subjects must have 20/40 (corrected) vision. Subjects who are blind cannot participate.

Day of testing eligibility

* Subjects must not have consumed caffeine within the last 12 hours
* Subjects must have slept >2 hours of their normal reported sleep time .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Profile of Moods Survey (POMS) Fatigue | change in fatigue from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  0-20 scale with higher scores being worse outcome
Profile of Moods Survey (POMS) Vigor | change in vigor from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  0-20 scale with higher scores being better outcome
Profile of Moods Survey (POMS) Tension | change in tension from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  0 to 20 scale with higher scores being worse outcome
Profile of Moods Survey (POMS) Depression | change in depression from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  0 to 20 scale with higher scores being worse outcome
Profile of Moods Survey (POMS) Anger | change in anger from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  0 to 20 scale with higher scores being worse outcome
Profile of Moods Survey (POMS) Confusion | change in confusion from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  -4 to 16 scale with higher scores being worse outcome
Profile of Moods Survey (POMS) Total Mood Disturbance | change in total mood disturbance from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  -24 to 96 with higher scores being worse outcomes
State Mental Energy | change in state mental energy from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  0 to 300 with higher scores being better outcomes
State Physical Energy | change in state physical energy from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  0 to 300 with higher scores being better outcomes
State Mental Fatigue | change in state mental fatigue from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  0 to 300 with higher scores being worse outcomes
State Physical Fatigue | change in state physical fatigue from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  0 to 300 with higher scores being worse outcomes
Gait speed | change in gait speed from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  gait speed in meters/second
Gait variability | change in variability from baseline to 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes during walking
  Variability in gait speed (reported as percent)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Boolani, PhD, Principal Investigator — Clarkson University
Locations (1):
- Clarkson University, Potsdam, New York, United States

IPD SHARING:
Plan to Share IPD: No